CLINICAL TRIAL: NCT05354102
Title: A Phase 1, Open-label Study to Evaluate the Safety and Tolerability of BMC128 in Combination With Nivolumab in Patients With Non-small Cell Lung Cancer (NSCLC), Melanoma or Renal Cell Carcinoma (RCC)
Brief Title: A First-in-human (FIH) Combination Treatment Study With a Single Dose Level of BMC128
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biomica Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMC128-001
Record Dates: First submitted 2022-04-20; First posted 2022-04-29 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Non-small Cell Lung Cancer; Melanoma; Renal Cell Carcinoma
Keywords: Microbiome
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Carcinoma, Renal Cell | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: One dose level of BMC128 will be investigated in combination with Nivolumab using a 3+3 model (Part A), followed by an expansion cohort (part B)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BMC128 in combination with Nivolumab (Experimental): Four 28-day treatment cycles of the standard Nivolumab treatment protocol (480 mg on Day 1 of each cycle) together with a QD regimen of BMC128, followed by a Iong-term Nivolumab monotherapy.
  Prior to starting this combination treatment, patients will undergo:
  I. Native microbiota depletion stage - patients will be treated with oral Vancomycin 500mg in combination with Neomycin 1000mg, q6h for 72 hours.
  II. BMC128 monotherapy induction stage - One BMC128 capsule will be administered once daily QD for a period of 14 days.
  Interventions: Drug: BMC128; Drug: Nivolumab

INTERVENTIONS:
Drug: BMC128 — A live bio-therapeutic product composed of 4 commensal bacterial strains, natural inhabitants of the human intestinal tract.
  Other Names: LBP (Live Bacteria Product)
Drug: Nivolumab — A human monoclonal antibody that blocks programmed-death-1 (PD-1). It is a type of immunotherapy and works as a checkpoint inhibitor, blocking a signal that prevents activation of T cells from attacking the cancer.
  Other Names: Opdivo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of BMC128 in combination with nivolumab (a known immunotherapy) in order to investigate if administration of select elements of the intestinal microbiome may serve as a novel and effective means of improving the efficacy of anti-cancer immunotherapies.

DETAILED DESCRIPTION:
This phase 1, first-in-human, proof-of-concept, open-label, combination treatment study is designed to profile the safety and tolerability of BMC128 in combination with Nivolumab, its effect on the intestinal microbiome and the anti-tumor immune and inflammatory responses and its preliminary anti-tumor activity. A 14-day induction phase, in which patients will be treated with a single dose level of BMC128, will be initiated, followed by four 28-day treatment cycles of BMC128 in combination with Nivolumab. Thereafter, patients will be treated with Nivolumab as a monotherapy for up to 22 additional cycles, until disease progression (PD) or intolerable toxicity

ELIGIBILITY:
Inclusion Criteria:

1. Capable of providing signed informed consent to participate in the study, and to comply with the requirements and restrictions listed in the protocol.
2. ≥18 years of age at time of informed consent
3. Histologically or cytologically confirmed metastatic or locally advanced unresectable clear cell renal cell carcinoma (ccRCC), cutaneous melanoma, or EGFR/ ALK wildtype adenocarcinoma-type non-small cell lung carcinoma (NSCLC).
4. At least one measurable lesion per RECIST v 1.1 criteria
5. Subjects must have progressed on treatment with a PD-1/PD-L1 inhibitor administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies. PD-1/PDL-1 inhibitor treatment progression is defined by meeting all of the following criteria:

   1. Has received at least 2 doses of a PD-1/PD-L1 inhibitor.
   2. Has demonstrated disease progression after PD-1/PD-L1 therapy as defined by RECIST v1.1, iRECIST or irRECIST. The initial evidence of disease progression (PD) is to be confirmed by a second assessment no less than four weeks from the date of the first documented PD, in the absence of rapid clinical progression.
   3. Progressive disease has been documented within 12 weeks from the last dose of a PD-1/PD-L1 inhibitor.
6. Subjects must have had prior response to anti-PD1/PDL-1 as single agent or in combination with other cancer therapies, defined as at least stable disease per iRECIST, as assessed by 2 consecutive imaging ≥ 4 weeks apart, with the first one performed no earlier than 9 weeks from initiation of anti PD1/PDL-1 treatment.
7. Subjects must demonstrate adequate organ functions at Screening:

   1. Absolute neutrophil count ≥1500/μL, platelet count ≥100,000/μL; hemoglobin ≥9.0 g/dL Note: Patients must not have received any growth factors or blood transfusions within 28 days prior to the Screening hematologic laboratory tests
   2. Total bilirubin <1.5 × the upper limit of normal (ULN) (with the exception of patients diagnosed with Gilbert syndrome), Alanine aminotransferase or aspartate aminotransferase <1.5 × ULN
   3. Creatinine ≤ 1.5 ULN and/or estimated glomerular filtration rate ≥ 60
   4. Albumin >30 g/L (3.0 g/dL)
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
9. Female subjects of childbearing potential should have a negative urine pregnancy test within 72 hours prior to enrolment (enrolment = start of depletion phase). If urine pregnancy results cannot be confirmed as negative, a SERUM β-HCG pregnancy test is required. Subjects of childbearing potential are those who have not been surgically sterilized or those age < 60 y who have not been free from menses for ≥2 years.
10. Female subjects of childbearing potential must be willing to use 2 methods of birth control starting from the start of the induction phase or be surgically sterile, or abstain from heterosexual activity throughout the course of the study and 120 days after the last dose of study medication
11. Male subjects with female partners of childbearing potential should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. History of partial or complete colon resection or colonic dissemination of tumor.
2. Active brain metastases or leptomeningeal disease. Subjects with asymptomatic central nervous system (CNS) metastases which have been stable (defined as without evidence of progression by magnetic resonance imaging (MRI) for at least 42 days prior to enrolment (initiation of depletion phase) and any neurologic symptoms have returned to baseline) following treatment with surgery or radiation therapy are allowed.
3. Prior solid organ or hematologic transplant.
4. Prior treatment with PD1/ PDL-1 inhibitor in combination with an immune-modifying microbiome agent.
5. History of treatment-related immune-mediated (or immune-related) adverse reactions to immune-modulatory agents (including but not limited to anti-PD1/PD-L1 agents, anti-CTLA4 monoclonal antibodies) that caused permanent discontinuation of the agent, or that were grade 3 or 4 in severity. Subjects with grade 3-4 hypothyroidism, primary adrenal insufficiency or diabetes mellitus which are asymptomatic following adequate supplementation, will be eligible.
6. Treatment with chemotherapy, immunotherapy, biologic therapy (except for denosumab and bisphosphonates), or other investigational agents <21 days of enrolment (initiation of depletion phase)
7. Palliative radiotherapy within 14 days or less from enrolment.
8. Comorbidity requiring corticosteroid therapy (>10mg prednisone/day or equivalent) within 7 days of enrolment. Physiologic replacement doses are allowed if they are ≤10mg of prednisone/day or equivalent, as long as they are not being administered for immunosuppressive intent. Inhaled, intranasal or topical steroids are permitted, provided that they are not for treatment of an autoimmune disorder.
9. Significant cardiac disease; New York Heart Association classification for chronic heart failure III-IV, symptomatic coronary artery disease, significant ventricular arrhythmias, myocardial infarction within 6 months, unstable, poorly controlled angina pectoris
10. Active, known or suspected autoimmune disease that has required systemic treatment within the past 2 years (i.e., with use of disease-modifying agents, corticosteroids or immunosuppressive drugs), except for replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.).

    Note: corticosteroids given within 24 hours of an imaging study for purposes of pre-medication in subjects with hypersensitivity to radiologic contrast agents are allowed
11. Serious active infection requiring systemic therapy
12. Subject has completed a course of antibiotics within the four weeks prior to enrollment
13. Subjects, who, in the opinion of the investigator, have predisposing risk factors for recurrent infections requiring systemic antibiotic treatment (i.e., fistulae, obstructing pulmonary mass, non-healing wound)
14. A known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the trial
15. Receipt of a live-virus vaccination within 28 days of enrolment. COVID-19 vaccine is not mandatory. However, patients who have been vaccinated against COVID-19 prior to study entry, should have completed the primary series of vaccination (initial two doses of the vaccine) at least 3 days before enrolment.
16. Known HIV infection, or active infection with hepatitis B or C
17. History of (non-infectious) pneumonitis that required steroids or has current active pneumonitis
18. Known additional malignancy either progressing or requiring active treatment (except for non-melanoma skin cancer, in situ cervical cancer or prostate intraepithelial neoplasia) within the last 2 years.
19. Female subjects who are breastfeeding
20. Known intolerance or hypersensitivity to study drugs
21. Known intolerance or hypersensitivity to oral vancomycin or neomycin
22. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
23. Known inability to orally ingest capsules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number and severity of drug-related treatment emergent adverse events (TEAEs) | Through study completion, an average of 1 year
  Safety and tolerability assessments will be based on frequency, severity, and duration of treatment-related AEs, including clinically significant changes from baseline in physical examination findings, vital signs, ECOG, and safety laboratory tests. All treatment-emergent adverse events (TEAEs) will be graded using NCI Common Terminology Criteria for Adverse Events 5.0 (CTCAE 5.0 or higher).

OTHER OUTCOMES:
The clinical effects of combined BMC128 and nivolumab treatment | Through study completion, an average of 1 year
  Objective response rate (ORR) defined as the proportion of patients who achieved partial response (PR) and complete response (CR), per iRECIST.
  Clinical benefit rate (CBR), defined as the proportion of patients who achieved PR, CR or stable disease (SD) for 6 months or more, per iRECIST.
  Duration of response (DoR) defined as time from response to progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Perets, Dr., Principal Investigator — Rambam MC
Locations (1):
- Rambam MC, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No